CLINICAL TRIAL: NCT00728117
Title: Should Very Low Birth Weight Infants Receive Enteral Nutrition During Indomethacin or Ibuprofen Treatment of a Patent Ductus Arteriosus? A Multi-Center Randomized Controlled Trial
Brief Title: Feeding During Ibuprofen or Indomethacin Treatment of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC3
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Patent Ductus Arteriosus
Keywords: indomethacin; ibuprofen; preterm infant
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ibuprofen-feeding (Experimental): Study infants will receive trophic enteral nutrition (15 ml/kg/day) during the study drug period.The study drug period is defined as the interval between administration of the first dose of ibuprofen and 24 hours after the last dose of ibuprofen.
  Interventions: Other: feeding
- ibuprofen-fasting (Experimental): Study infants will be fasted during the study drug period.The study drug period is defined as the interval between administration of the first dose of ibuprofen and 24 hours after the last dose of ibuprofen.
  Interventions: Other: fasting
- indomethacin-feeding (Experimental): Study infants will receive trophic enteral nutrition (15 ml/kg/day) during the study drug period.The study drug period is defined as the interval between administration of the first dose of indomethacin and 24 hours after the last dose of indomethacin.
  Interventions: Other: feeding
- indomethacin-fasting (Experimental): Study infants will be fasted during the study drug period.The study drug period is defined as the interval between administration of the first dose of indomethacin and 24 hours after the last dose of indomethacin.
  Interventions: Other: fasting

INTERVENTIONS:
Other: feeding — Study infants will receive trophic enteral nutrition (15 ml/kg/day) during the study drug period.The study drug period is defined as the interval between administration of the first dose of ibuprofen or indomethacin and 24 hours after the last dose of ibuprofen or indomethacin.
  Arms: ibuprofen-feeding; indomethacin-feeding
Other: fasting — Study infants will be fasted during the study drug period.The study drug period is defined as the interval between administration of the first dose of ibuprofen or indomethacin and 24 hours after the last dose of ibuprofen or indomethacin.
  Arms: ibuprofen-fasting; indomethacin-fasting

SUMMARY:
We hypothesize that feeding preterm infants while they receive indomethacin or ibuprofen therapy for treatment of a patent ductus arteriosus will decrease the incidence of feeding intolerance and shorten the time period that infants need to tolerate full enteral nutrition. We also hypothesize that this intervention will minimize the alterations in intestinal permeability that occur with these drugs and will improve the infants' hemodynamic response to enteral nutrition

DETAILED DESCRIPTION:
This study is a randomized controlled multi-center clinical trial to determine whether very low birth weight infants should receive feedings during indomethacin or ibuprofen treatment of a patent ductus arteriosus (PDA). Many neonatologists withhold feeds from premature infants receiving indomethacin or ibuprofen therapy for a PDA because of concerns that these drugs alter intestinal blood flow and permeability. However, there are no established studies which show that feeding during these medical treatments leads to bowel injury. At the same time, studies suggest that withholding feedings from premature infants may lead to intestinal atrophy and injury, leading to increased difficulty with feedings when they are initiated or re-started. Thus, this multi-center study evaluates whether feeding infants during indomethacin or ibuprofen therapy improves feeding tolerance by measuring the number of episodes of feeding intolerance and the number of days required to attain full feedings. In addition, this study will employ techniques to measure gastrointestinal permeability and mesenteric blood flow in patients who receive and don't receive feedings for their PDA treatment.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 401-1,250 g birth weight who

  * Are receiving or are scheduled to begin enteral feedings and
  * Are about to receive pharmacologic treatment (either indomethacin or ibuprofen) to close their PDA.

Exclusion Criteria:

* Serious congenital malformations
* Chromosomal anomalies
* Congenital or acquired gastrointestinal anomalies
* Prior episode of necrotizing enterocolitis
* Use of inotropic support for hypotension
* Renal anomalies or disease
* Are receiving > 80 ml/kg/d of enteral feeding

Ages: 23 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Assess the effect of feeding infants during indomethacin or ibuprofen therapy on the incidence of feeding intolerance and the number of days required to achieve full feedings (120 ml/kg/day). | 4 years

SECONDARY OUTCOMES:
incidence of necrotizing enterocolitis or spontaneous perforation | 4 years
Assess the effect of feeding very low birth weight infants during indomethacin or ibuprofen therapy on intestinal permeability. | 4 years
Assess the effect of feeding very low birth weight infants during indomethacin or ibuprofen therapy on the normal hyperemic response to feeding. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Clyman, M.D., Principal Investigator — University of California, San Francisco
Locations (14):
- United States (14):
  - University of California san Francisco, San Francisco, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Children's Memorial Hospital-Northwestern University, Chicago, Illinois
  - North Shore University Health System, Northwestern University, Evanston, Illinois
  - Boston University-Boston Medical Center, Boston, Massachusetts
  - Children's Hospital-Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Children's Hospital-Saint Paul, Saint Paul, Minnesota
  - Atlantic Health Organization, Morristown, New Jersey
  - Columbia University, New York, New York
  - Case Western Reserve, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Virginia, Charlottesville, Charlottesville, Virginia

REFERENCES:
- [Derived] Yanowitz TD, Reese J, Gillam-Krakauer M, Cochran CM, Jegatheesan P, Lau J, Tran VT, Walsh M, Carey WA, Fujii A, Fabio A, Clyman R. Superior mesenteric artery blood flow velocities following medical treatment of a patent ductus arteriosus. J Pediatr. 2014 Mar;164(3):661-3. doi: 10.1016/j.jpeds.2013.11.002. Epub 2013 Dec 8. PMID 24321538
- [Derived] Clyman R, Wickremasinghe A, Jhaveri N, Hassinger DC, Attridge JT, Sanocka U, Polin R, Gillam-Krakauer M, Reese J, Mammel M, Couser R, Mulrooney N, Yanowitz TD, Derrick M, Jegatheesan P, Walsh M, Fujii A, Porta N, Carey WA, Swanson JR; Ductus Arteriosus Feed or Fast with Indomethacin or Ibuprofen (DAFFII) Investigators. Enteral feeding during indomethacin and ibuprofen treatment of a patent ductus arteriosus. J Pediatr. 2013 Aug;163(2):406-11. doi: 10.1016/j.jpeds.2013.01.057. Epub 2013 Mar 6. PMID 23472765